CLINICAL TRIAL: NCT02100046
Title: Assessment of the Effectiveness of Ethosuximide in the Treatment of Peripheral Neuropathic Pain.
Acronym: EDONOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0186; 2013-004801-26
Record Dates: First submitted 2014-03-20; First posted 2014-03-31 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Neuropathic Traumatic Pain; Pain NRS ≥ 4; Peripheral Neuropathic Pain; Neuropathic Pain Diagnostic Questionnaire (DN4) ≥ 4
Keywords: Ethosuximide; Neuropathic pain; Pain; Quality of life; Neuropathic Pain diagnostic questionnaire ≥ 4; Analgesic treatment failure for at least 3 months
MeSH Terms: conditions — Neuralgia; Pain | interventions — Ethosuximide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ethosuximide (Experimental): The purpose of this study is to assess the effectiveness of ethosuximide (Zarontin®) on the pain symptoms and quality of life in patients with neuropathic traumatic pain compared to a control group.
  Interventions: Drug: Zarontin® (ethosuximide) and Stodal®
- control group (Other): The purpose of this study is to assess the effectiveness of ethosuximide (Zarontin®) on the pain symptoms and quality of life in patients with neuropathic traumatic pain compared to a control group.
  Interventions: Drug: Zarontin® (ethosuximide) and Stodal®

INTERVENTIONS:
Drug: Zarontin® (ethosuximide) and Stodal®
  Other Names: Zarontin® (ethosuximide), administration: oral syrup using a graduated pipette. Duration of treatment: 42 days; Inactive substance: Stodal® administration: oral syrup using a graduated pipette. Duration of treatment: 42 days. Same dosage as Zarontin®

SUMMARY:
Currently, it is established that the voltage-gated calcium channels modulate pain perception due to an influence on the neuronal transmission and excitability. In the past, attention has focused on the modulation of high voltage activated calcium channel. More recently, scientific interest has proven to the low voltage activated calcium channel, also called T-type channels. The data from the literature show significant involvement of these channels in the physiology of nociception and pathophysiology of acute and chronic pain. Moreover, in several animal pain models (acute, neuropathic, inflammatory), T-type channels inhibition alleviates painful behaviours.

Analgesics treatments available in clinic are ineffective in some patients with chronic pain (neuropathic, inflammatory) and often induce deleterious side effects. Thus, the clinical use of selective inhibitors of T-type channels could not only help the development of new therapies for the treatment of neuropathic pain (prevalence = 5-8 %), but also have a pharmaco-economic impact due to the low selling price of their inhibitor currently available: Zarontin®.

The purpose of this study is to assess the effectiveness of ethosuximide (Zarontin®) on the pain symptoms and quality of life in patients with peripheral neuropathic pain compared to a control group.

DETAILED DESCRIPTION:
This is a multicentre, parallel-group, double-blind, randomised clinical trial comparing ethosuximide and inactive control for the treatment of peripheral neuropathic pain, assessed by numerical rating scale and quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Traumatic neuropathy or post-surgical (excluding amputations) with Neuropathic -Pain Diagnostic DN4 ≥ 4 positive and IASP criteria
* ENS pain ≥ 4
* ALT, AST, PAL, normal GGT, creatinine <133μmol / L, hematocrit> 38%, β-HCG
* Patients affiliated to the French Social Security
* Patients with free and informed consent has been obtained
* Peripheral neuropathic pain with Neuropathic Pain Diagnostic DN4 ≥ 4 positive

Exclusion Criteria:

* Pregnancy or breastfeeding
* Diabetic neuropathy, post-herpetic neuralgia, cancer or chemotherapy-induced,
* Patients with impaired glucose tolerance,
* Medical and surgical history incompatible with the study,
* History of renal disease and / or liver,
* Addiction to alcohol and / or drugs,
* Taking antiepileptic family carboxamides and ethosuximide
* Use of St. John's wort,
* Allergy succinimides (ethosuximide, methsuximide, phensuximide)
* Psychotic disorders,
* Patients with epilepsy,
* Patient exclusion period, or the total allowable compensation exceeded
* Patients undergoing a measure of legal protection (guardianship, supervision ...)
* Central neuropathic pain
* Other chronic pain (osteoarthritis, arthritis, fibromyalgia…) with intensity greater than neuropathic pain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the analgesic efficacy of ethosuximide in peripheral neuropathic pain patients | day 43
  Δ = score NRS (Day 0) - score NRS (D +43)

SECONDARY OUTCOMES:
Impact of ethosuximide on neuropathic pain | after day 43
Quality of life | after day 43
sleep and the overall impression of patients | after day 43

CONTACTS AND LOCATIONS:
Overall Officials: Alain ESCHALIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Kerckhove N, Pereira B, Soriot-Thomas S, Alchaar H, Deleens R, Hieng VS, Serra E, Lanteri-Minet M, Arcagni P, Picard P, Lefebvre-Kuntz D, Maindet C, Mick G, Balp L, Lucas C, Creach C, Letellier M, Martinez V, Navez M, Delbrouck D, Kuhn E, Piquet E, Bozzolo E, Brosse C, Lietar B, Marcaillou F, Hamdani A, Leroux-Bromberg N, Perier Y, Vergne-Salle P, Gov C, Delage N, Gillet D, Romettino S, Richard D, Mallet C, Bernard L, Lambert C, Dubray C, Duale C, Eschalier A. Efficacy and safety of a T-type calcium channel blocker in patients with neuropathic pain: A proof-of-concept, randomized, double-blind and controlled trial. Eur J Pain. 2018 Aug;22(7):1321-1330. doi: 10.1002/ejp.1221. Epub 2018 Apr 18. PMID 29577519
- [Derived] Kerckhove N, Mallet C, Pereira B, Chenaf C, Duale C, Dubray C, Eschalier A. Assessment of the effectiveness and safety of Ethosuximide in the Treatment of non-Diabetic Peripheral Neuropathic Pain: EDONOT-protocol of a randomised, parallel, controlled, double-blinded and multicentre clinical trial. BMJ Open. 2016 Dec 16;6(12):e013530. doi: 10.1136/bmjopen-2016-013530. PMID 27986742